PRoVENT-IMIC: Statistical Analysis Plan

updated 20 Dic 2018

confidence levels.

General description of statistical methods

Normally distributed variables will be expressed by their mean and standard deviation; not normally distributed variables will be expressed by their medians and interquartile ranges; categorical variables will be expressed as n (%). In test groups of continuous normally distributed variables, Student's t-test will be used. Likewise if continuous data are not normally distributed the Mann Whitney U test will be used. Categorical variables will be compared with the Chi-square test or Fisher's exact test or when appropriate as relative risks. Statistical uncertainty will be expressed by 95%

Time to ICU discharge will be analysed as a time to event variable using Cox proportional hazard models and visualized by Kaplan–Meier curves. Time–course variables (e.g. repeated measures of ventilatory parameters, vital signs, oxygenation parameters and others) will be analysed using mixed–effect longitudinal models with random intercepts for patients and centers; time will be treated as a continuous variable. Multiple imputation of missing values will be considered when appropriate. No correction for multiple comparisons are pre-specified, thus, all the findings should be viewed as exploratory. Statistical analyses will be conducted using R (www.r-project.org). A *P*–value of less than 0.05 will be considered statistically significant.

Baseline descriptive statistics

Patients baseline characteristics will be presented as shown in **dummy Table 1.** The predicted bodyweight of male patients will be calculated as 50+0.91(height [cm]-152.4) and for female patients as 45.5+0.91(height [cm]-152.4). Patients will be grouped based on the risk of ARDS defined as a Lung injury prediction score (LIPS) equal or greater than 4.

Analysis of the primary outcome

The primary outcomes ( $V_T$  size [ml/kg PBW] and PEEP [cm  $H_2O$ ] levels during the first three days of mechanical ventilation), alike other ventilator settings – will be reported as in **dummy Table 2.** Variables that were collected daily (e.g. ventilator

1

parameters, respiratory rates, SpO2) will be presented as median [IQR]. They will be analysed and compared between patients at no risk for ARDS, patients at risk for ARDS and in patients with ARDS (in case the diagnosis of ARDS could be made on admission). Also, the ventilatory variables over the first three days will be presented in line plots and the *p* value will be calculated using mixed–effect longitudinal models with random intercepts for patients and centers and an interaction between time and the risk for ARDS as fixed effect; time will be treated as a continuous variable.

Scatterplots will be used to present distributions of  $V_T$  versus PEEP,  $V_T$  versus respiratory rate,  $V_T$  versus plateau pressure and  $V_T$  versus driving pressure. Cut-offs to form matrices will be based on widely accepted values for each variable, specifically 8 ml/kg PBW for  $V_T$ , 14 breaths per minute for respiratory rate, 30 cmH2O for plateau pressure, 5 cmH20 for PEEP and 15 cmH2O for driving pressure. Driving pressure will be calculated by subtracting the level of PEEP from the plateau pressure (Pplat in volume–control ventilation) or maximal airway pressure (Pmax in pressure–control ventilation).

## Analysis of the secondary outcomes

The number of patients developing a pulmonary complication during the first 7 days (excluding first day of mechanical ventilation) and patient outcomes at ICU discharge will be reported in absolute numbers and percentages (**dummy Table 3**).

Univariate analysis will be performed to identify potential factors associated with ICU mortality and development of pulmonary complications including, but not limited to, ventilator settings (in particular  $V_T$  and PEEP at day 0). Relevant covariates included in the final mixed-effect multivariable model will be identified as those with p < 0.2 in the univariable model (including participating center as a random effect), those with clinical relevance and without statistical association with other relevant variables. The linearity of each continuous predictor with the log odds outcome will be checked graphically and, if not present, a log-transformation will be performed. Pearson correlation coefficients will be used to assess collinearity between predictors. Since a high collinearity between peak, plateau and driving pressure is expected, the main model will consider the variable with the higher amount of measurements between peak or plateau pressure. Driving pressure will be considered in a sensitivity analysis, excluding PEEP, peak and plateau pressure. Finally, the intraclass correlation coefficient (ICC) will be assessed. The ICC

represents the ratio of between-site variance to total variance, ranging from 0 to 1.

Potential associations between ventilator settings and outcome will be explored in pre–specified subgroups by building a model in each category. The subgroups are: (1) patients at low risk of ARDS versus patients at risk of ARDS; (2) patients without ARDS versus patients with ARDS; (3) reason for ICU admission and (4) reason for start of invasive ventilation.

## Supplementary information

 Participant ICU structure and organizational descriptives will be reported in supplementary dummy Table 1, aggregated per country.

## **Dummy Table 1. Baseline patient characteristics**

| | All patients (n=) | At risk of ARDS | Not at risk of P- | |
|---|---|---|---|---|
| Ame (weeks) | mean ±SD or | (n=)<br>mean ±SD or | ARDS (n=) value mean ±SD or | le |
| Age (years) | median [IQR] | median [IQR] | median [IQR] | |
| Sex | median [iQit] | median [iQit] | median [iQit] | |
| female | n/total (%) | n/total (%) | n/total (%) | |
| Country | Tirtotal (70) | Tirtotal (70) | Tirtotai (70) | |
| Thailand | n/total (%) | n/total (%) | n/total (%) | |
| Vietnam | n/total (%) | n/total (%) | n/total (%) | |
| Sri Lanka | n/total (%) | n/total (%) | n/total (%) | |
| Maldives | n/total (%) | n/total (%) | n/total (%) | |
| Bangladesh | n/total (%) | n/total (%) | n/total (%) | |
| Pakistan | n/total (%) | n/total (%) | n/total (%) | |
| India | n/total (%) | n/total (%) | n/total (%) | |
| Malaysia | n/total (%) | n/total (%) | n/total (%) | |
| Myanmar | n/total (%) | n/total (%) | n/total (%) | |
| Iran | n/total (%) | n/total (%) | n/total (%) | |
| Nepal | n/total (%) | n/total (%) | n/total (%) | |
| Severity of illness, SOFA score | | | | |
| Total | median [IQR] | median [IQR] | median [IQR] | |
| Pulmonary | median [IQR] | median [IQR] | median [IQR] | |
| Haematological | median [IQR] | median [IQR] | median [IQR] | |
| Liver | median [IQR] | median [IQR] | median [IQR] | |
| Circulation | median [IQR] | median [IQR] | median [IQR] | |
| Neurology<br>Renal | median [IQR]<br>median [IQR] | median [IQR]<br>median [IQR] | median [IQR]<br>median [IQR] | |
| LIPS | mean ±SD or | mean ±SD or | mean ±SD or | |
| LIFS | median [IQR] | median [IQR] | median [IQR] | |
| Body mass index (kg/m²) | mean ±SD or | mean ±SD or | mean ±SD or | |
| , , , | median [IQR] | median [IQR] | median [IQR] | |
| Predicted body weigth (kg) | mean ±SD or | mean ±SD or | mean ±SD or | |
| | median [IQR] | median [IQR] | median [IQR] | |
| Smoker | n/total (%) | n/total (%) | n/total (%) | |
| Never | n/total (%) | n/total (%) | n/total (%) | |
| Former | n/total (%) | n/total (%) | n/total (%) | |
| Current | n/total (%) | n/total (%) | n/total (%) | |
| Unknown Reason for ICU admission | n/total (%) | n/total (%) | n/total (%) | |
| | - /t - t - 1 (O/) | /t - t - L /O/ \ | - 4-1-1 (0/) | |
| Planned surgery | n/total (%) | n/total (%) | n/total (%) | |
| Emergency Surgery (excluding trauma) Trauma | n/total (%)<br>n/total (%) | n/total (%)<br>n/total (%) | n/total (%)<br>n/total (%) | |
| Medical condition | n/total (%) | n/total (%) | n/total (%) | |
| Non invasive ventilation before intubation | n/total (%) | n/total (%) | n/total (%) | |
| Duration (minutes) | mean ±SD or | mean ±SD or | mean ±SD or | |
| Burdion (minutes) | median [IQR] | median [IQR] | median [IQR] | |
| Invasive ventilation in the ward for > 12h | n/total (%) | n/total (%) | n/total (%) | |
| before ICU admission | . , | . , | ` , | |
| High risk surgery | n/total (%) | n/total (%) | n/total (%) | |
| Admission source | | | | |
| Emergency department | n/total (%) | n/total (%) | n/total (%) | |
| Operating room | n/total (%) | n/total (%) | n/total (%) | |
| Ward | n/total (%) | n/total (%) | n/total (%) | |
| Directly from community | n/total (%) | n/total (%) | n/total (%) | |
| Reason for intubation | . , | . , | · / | |
| Cardiac arrest | n/total (%) | n/total (%) | n/total (%) | |
| Anesthesia for surgery (planned) | n/total (%) | n/total (%) | n/total (%) | |
| Depressed level of consciousness | n/total (%) | n/total (%) | n/total (%) | |
| Acute respiratory failure | n/total (%) | n/total (%) | n/total (%) | |
| Hemodynamic instability | n/total (%) | n/total (%) | n/total (%) | |
| Other | n/total (%) | n/total (%) | n/total (%) | |
| Cause of Acute Respiratory Failure | | | | |
| Community acquired pneumonia | n/total (%) | n/total (%) | n/total (%) | _ |
| Nosocomial pneumonia | n/total (%) | n/total (%) | n/total (%) | |
| Unplanned post operative ventilation | n/total (%) | n/total (%) | n/total (%) | |
| Cardiogenic pulmonary edema | n/total (%) | n/total (%) | n/total (%) | |

| Sepsis (other than pneumonia) | n/total (%) | n/total (%) | n/total (%) |
|-------------------------------|-------------|-------------|-------------|
| COPD exacerbation | n/total (%) | n/total (%) | n/total (%) |
| ARDS | n/total (%) | n/total (%) | n/total (%) |
| Other | n/total (%) | n/total (%) | n/total (%) |
| Chronic comorbidity | | | |
| None | n/total (%) | n/total (%) | n/total (%) |
| Arterial hypertension | n/total (%) | n/total (%) | n/total (%) |
| Heart Failure | n/total (%) | n/total (%) | n/total (%) |
| Diabetes Mellitus | n/total (%) | n/total (%) | n/total (%) |
| Chronic Kidney Disease | n/total (%) | n/total (%) | n/total (%) |
| Liver Cirrhosis | n/total (%) | n/total (%) | n/total (%) |
| COPD | n/total (%) | n/total (%) | n/total (%) |
| Cancer | n/total (%) | n/total (%) | n/total (%) |
| Neuromuscular disease | n/total (%) | n/total (%) | n/total (%) |
| Other | n/total (%) | n/total (%) | n/total (%) |

Dummy Table 2. Ventilation characteristics in first 3 days of mechanical ventilation

| | | Day 0 | | | Day 01 | | | Day 02 | | | Day 03 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | At Risk | Not At<br>Risk | p value | At Risk | Not At<br>Risk | p value | At Risk | Not At<br>Risk | p value | At Risk | Not At<br>Risk | p value |
| Absolute V <sub>⊤</sub> | median | | | | | | | | | | | |
| V <sub>⊤</sub> (ml/kg PBW) | median | | | | | | | | | | | |
| Controlled ventilation mode | median | | | | | | | | | | | |
| Spontaneous ventilation mode | median | | | | | | | | | | | |
| V <sub>T</sub> ≤7 | n/total (%) | | | | | | | | | | | |
| V <sub>7</sub> 7–8 | n/total (%) | | | | | | | | | | | |
| V <sub>7</sub> 9–10 | n/total (%) | | | | | | | | | | | |
| V <sub>7</sub> ≥ 10 | n/total (%) | | | | | | | | | | | |
| PEEP (cm H <sub>2</sub> O) | mean ±SD | | | | | | | | | | | |
| N 55 | n/total (%) | | | | | | | | | | | |
| 8-9 | n/total (%) | | | | | | | | | | | |
| 9–10 | n/total (%) | | | | | | | | | | | |
| ≥10 | n/total (%) | | | | | | | | | | | |
| Mode of Ventilation | | | | | | | | | | | | |
| Volume-controlled | n/total (%) | | | | | | | | | | | |
| Pressure-controlled | n/total (%) | | | | | | | | | | | |
| PSV | n/total (%) | | | | | | | | | | | |
| SIMV | n/total (%) | | | | | | | | | | | |
| APRV | n/total (%) | | | | | | | | | | | |
| Other | n/total (%) | | | | | | | | | | | |
| Peak pressure (cm H <sub>2</sub> O) | median | | | | | | | | | | | |
| Plateau pressure (cm H <sub>2</sub> O) | median | | | | | | | | | | | |
| Number of patients | median | | | | | | | | | | | |
| Driving pressure | median | | | | | | | | | | | |
| Static compliance (ml/cmH2O) | median | | | | | | | | | | | |
| Respiratory rate (breaths per | median | | | | | | | | | | | |
| Fi02 | median | | | | | | | | | | | |
| Minute Ventilation (L/min) | median | | | | | | | | | | | |
| PaO <sub>2</sub> /FiO <sub>2</sub> | median | | | | | | | | | | | |
| SpO <sub>2</sub> /FiO <sub>2</sub> | median | | | | | | | | | | | |
| PaCO <sub>2</sub> | median | | | | | | | | | | | |
| Arterial blood pH | median | | | | | | | | | | | |
| HCO <sub>3</sub> (mEq/L) | median | | | | | | | | | | | |
| Arterial lactate levels (meq/L) | median | | | | | | | | | | | |
| Use of neuromuscular blockers | n/total (%) | | | | | | | | | | | |
| Use of prone positioning | n/total (%) | | | | | | | | | | | |
| Use of recruitment manouvers | n/total (%) | | | | | | | | | | | |

Dummy Table 3. Pulmonary complications observed in first 7 days of MV and clinical outcomes

| Complication | All (n=) | At risk of ARDS (n=) | Not at risk (n=) |
|---|---|---|---|
| Any pulmonary complication | n/total (%) | | |
| Pulmonary infection | n/total (%) | | |
| confirmed by microbiology | n/total (%) | | |
| ARDS | n/total (%) | | |
| mild | n/total (%) | | |
| moderate | n/total (%) | | |
| severe | n/total (%) | | |
| Pneumothorax | n/total (%) | | |
| Pleural effusion | n/total (%) | | |
| Atelectasis | n/total (%) | | |
| Cardiogenic pulmonary edema | n/total (%) | | |
| New pulmonary infiltrates | n/total (%) | | |
| Outcome | | | |
| Death in ICU | n/total (%) | | |
| Transferred to ward | n/total (%) | | |
| Discharged home | n/total (%) | | |
| Transferred to other ICU | n/total (%) | | |
| Transferred to medium care or HDU | n/total (%) | | |
| Palliative care | n/total (%) | | |
| Duration of MV (days) | mean ±SD or median [IQR] | | |
| Length of stay in ICU | mean ±SD or median [IQR] | | |
| Tracheostomy | n/total (%) | | |

| _ |
|------------------------------------------|
| $\subseteq$ |
| 뒫 |
| $\subseteq$ |
| 3 |
| 0 |
| ပ |
| _ |
| Φ |
| ed per country |
| ~ |
| Š |
| aggregate |
| ā |
| 0 |
| Ō |
| ≦ |
| 0 |
| 0 |
| Ŋ |
| <u>.2</u> |
| Ŧ |
| <u>.s</u> |
| Ž |
| ā |
| ਹ |
| ă |
| Ξ |
| Ø |
| 드 |
| ပ |
| 'n |
| Ľ |
| ø |
| Ħ |
| $\overline{}$ |
| w |
| $\tilde{a}$ |
| Ö |
| Ω<br>Ω |
| ngc |
| ting c |
| ating c |
| pating c |
| sipating c |
| icipating c |
| rticipating c |
| articipating c |
| Participating c |
| . Participating centers characteristics, |
| Ć. |
| Ć. |
| Ć. |
| Ć. |
| Ć. |
| / Table 1. |
| / Table 1. |
| / Table 1. |
| / Table 1. |
| / Table 1. |
| / Table 1. |
| / Table 1. |
| Ć. |
| / Table 1. |

| Number of participating centers Hospital status n/total (%) Private n/total (%) Hospital type n/total (%) Academic n/total (%) Non-academic n/total (%) Non-academic n/total (%) Rural n/total (%) Mixed n/total (%) Surgical n/total (%) Medical n/total (%) Neurological n/total (%) Neurological n/total (%) | |
|---|---|
| lation served | I TOR! |
| lation served | |
| ic lation served | |
| c ation served | |
| | 1 IQRI |
| cic | 1 IQRI |
| cic | I IQRI |
| cic<br>-I | I IQRI |
| ojc<br> | I IQRI |
| cic<br> | I IQRI |
| भ।<br>thoracic<br>ogical | I IQRI |
| thoracic<br>ogical | I IQRI |
| ogical | I IQRI |
| • | I IQRI |
| Mixed | I IQRI |
| ICU arrangement | I IORI |
| Onen C | IOR |
| 7 | IORI |
| Total number of beds in Hospital mean ±SD or median [IQR] | |
| Number of beds in ICU mean ±SD or median [IQR] | l [IQR] |
| Total number of ICU admissions in 2017 mean ±SD or median IIQRI | IJORI |
| | 1 |
| Total number of ICU admissions during the mean ±SD or median [IQR] PRoVENT-iMIC study period (28 days) | [IQR] |
| ICUs involved in research activities n/total (%) | |
| Total number of mechanical ventilators in unit mean ±SD or median [IQR] | , flori |
| Number of functioning ventilators mean ±SD or median [IQR] | I [IQR] |
| Type of humidification mostly used Active humidification HME | |
| Routine use of Non Invasive Ventilation (NIV) n/total (%) | |
| Availability of high flow nasal oxygen (HFNT) n/total (%) devices? | |
| Dedicated physician available in ICU 24/7 n/total (%) | |
| Number of staff physicians per shift median [IQR] | |

| Country | Country1 | Country2 | Country10 |
|---|---|---|---|
| Number of doctors in training or residents per shift | median [IQR] | | |
| Number of Nurses per shift | median [IQR] | | |
| Usual nurse to bed ratio | | | |
| 1 nurse to 1 bed | n/total (%) | | |
| 1 nurse to 2 beds | n/total (%) | | |
| 1 nurse to 3 beds | n/total (%) | | |
| 1 nurse to 4 beds | n/total (%) | | |
| Other | n/total (%) | | |
| Availability of renal replacement therapy | n/total (%) | | |
| Availability of pulse oximetry for all patients | n/total (%) | | |
| Availability of end tidal CO <sub>2</sub> | n/total (%) | | |
| Availability of chest x-ray apparatus | | | |
| Not available | n/total (%) | | |
| Dedicated ICU portable apparatus | n/total (%) | | |
| Hospital apparatus | n/total (%) | | |
| External provider | n/total (%) | | |
| Availability of computed tomography imaging | | | |
| Not available | n/total (%) | | |
| In hospital | n/total (%) | | |
| Outsourced | n/total (%) | | |
| Availability of ultrasound apparatus | | | |
| Not available | n/total (%) | | |
| Yes, dedicated ICU ultrasound apparatus | n/total (%) | | |
| Yes, in hospital | n/total (%) | | |
| Availability of blood gas analyzer in ICU | n/total (%) | | |